CLINICAL TRIAL: NCT02997917
Title: Factors That Determine the Response to Meal Ingested: Education
Brief Title: Effect of Education on the Responses to Meal Ingestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PR(AG)338/2016A
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
MeSH Terms: interventions — Educational Status; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education (Experimental): Solutions of the five basic tastes (sweet, salty, sour, bitter and umami) and the 3 main components of the probe soup (onion, leek and carrot) will be given every 10 min with a mouthwash after each test. In the real education group, solutions at suprathreshold concentration for detection will be given with a subsequent comment on the flavor and an explanation of the components and preparation of the soup (low temperature cooking to preserve flavors).
  Interventions: Behavioral: Education
- Sham (Sham Comparator): Solutions of the five basic tastes (sweet, salty, sour, bitter and umami) and the 3 main components of the probe soup (onion, leek and carrot) will be given every 10 min with a mouthwash after each test. In the sham education group solutions at subthreshold concentration for detection with no explanation will be provided.
  Interventions: Behavioral: Sham

INTERVENTIONS:
Behavioral: Education
  Arms: Education
Behavioral: Sham
  Arms: Sham

SUMMARY:
The effect of education on the responses to a probe meal (250 mL vegetable soup cooked at low temperature and 25 g bread) will be studied in a parallel design. The effects of education will be tested in two different groups in random order: real versus sham education. In each group the responses to a probe meal will be tested on 2 different days before and after the intervention. Participants will be instructed to eat a standard dinner the day before, to consume a standard breakfast at home after overnight fast, and to report to the laboratory, where the probe meal will be administered 3 h after breakfast. Studies will be conducted in a quiet, isolated room with participants sitting on a chair. Perception will be measured at 5 min intervals 10 min before and 20 min after ingestion and at 10 min intervals up to 60 min after the probe meal.

ELIGIBILITY:
Inclusion Criteria:

- non-obese

Exclusion Criteria:

* history of gastrointestinal symptoms
* prior obesity
* use of medications
* history of anosmia and ageusia
* current dieting
* alcohol abuse
* psychological disorders
* eating disorders

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in digestive well-being measured after a test meal by the end of the intervention versus before. | 1 day
  Change in average well-being measured by 0-10 score scales at the end of the test meal administered before and after intervention.

SECONDARY OUTCOMES:
Change in satiety measured after a test meal by the end of the intervention versus before | 1 day
  Change in average satiety measured by 0-10 score scales at the end of the test meal administered before and after intervention.
Change in fullness sensation measured after a test meal by the end of the intervention versus before. | 1 day
  Change in average fullness measured by 0-10 score scales at the end of the test meal administered before and after intervention.
Change in discomfort/pain measured after a test meal by the end of the intervention versus before | 1 day
  Change in average fullness measured by 0-10 score scales at the end of the test meal administered before and after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Azpiroz, MD, Principal Investigator — University Hospital Vall d'Hebron
Locations (1):
- Fernando Azpiroz, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No